CLINICAL TRIAL: NCT04264156
Title: A Multinational, Multicenter, Masked, Randomized, Controlled Study to Assess the Safety and Efficacy of Lucinactant for Inhalation Versus nCPAP Alone in Preterm Neonates 26 to 32 Weeks Gestational Age With RDS
Brief Title: A Safety and Efficacy Study of Lucinactant for Inhalation in Preterm Neonates 26 to 32 Weeks Gestational Age
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Corporate business reasons
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-CL-1702
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: intubation; surfactant; continuous positive airway pressure; aerosol; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome | interventions — lucinactant; Inhalation

STUDY DESIGN:
Intervention Model Description: This study is a multinational, multicenter, double-blind (masked), parallel group, randomized, controlled study, in preterm neonates 26 to 32 completed weeks post-menstrual age (PMA).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The first 2 subjects at each site for each cohort will be dosed with open-label active treatment for training purposes. Following the first 2 subjects, preparation and delivery of treatment will be blinded from the study staff. Treatment will be delivered behind a partition and no information about treatment will be given to investigator, parents, or other applicable study staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Lucinactant (160 mg/kg) + nCPAP (Experimental): Lucinactant for inhalation, 160 mg total phospholipids (TPL)/kg Delivered as an aerosol once, with up to 3 repeats of 80 mg/kg allowed within 36 hours of birth
  Interventions: Combination Product: Lucinactant for Inhalation
- nCPAP Only (Sham Comparator): nCPAP Only as sham comparator. Bubble nCPAP is standard of care. Treatment time behind barrier to match active treatment delivery time
  Interventions: Other: nCPAP Only

INTERVENTIONS:
Combination Product: Lucinactant for Inhalation — A drug-device combination product that delivers aerosolized SRT to preterm neonates with RDS who are being supported with nasal continuous positive airway pressure (nCPAP).
  Other Names: AEROSURF
  Arms: Lucinactant (160 mg/kg) + nCPAP
Other: nCPAP Only — Nasal continuous positive airway pressure (nCPAP) alone
  Arms: nCPAP Only

SUMMARY:
This study is to evaluate the safety and efficacy of lucinactant for inhalation in conjunction with nCPAP, in comparison to nCPAP alone, in preterm neonates with RDS, as assessed by the incidence of and time to respiratory failure and/or death due to RDS in the first 72 hours and 28 days of life. Half of the subjects will receive lucinactant for inhalation and half will receive standard of care (nCPAP alone).

DETAILED DESCRIPTION:
An unmet medical need exists for a means to deliver surfactant replacement therapy (SRT) to preterm neonates with RDS supported with nCPAP early in the course of the disease. This strategy has the potential to improve RDS prior to the development of respiratory failure, thereby avoiding the need for endotracheal intubation and mechanical ventilation (MV), or reduce the duration of MV, and the resultant potential for morbidity and complications. The ability to administer SRT via aerosol has the potential to address this unmet need.

Lucinactant for inhalation (AEROSURF) is an investigational drug-device combination product, designed to deliver aerosolized SRT to preterm neonates with RDS who are being supported with nCPAP. The drug component of lucinactant for inhalation is lyophilized lucinactant, a lyophilized form of SURFAXIN® (lucinactant) Intratracheal Suspension. The device component, the AEROSURF Delivery System (ADS), the next-generation device following use of the prototype device in earlier trials, uses novel technology to aerosolize lucinactant for inhalation.

This study evaluates the safety and efficacy of lucinactant for inhalation in conjunction with nCPAP, in comparison to nCPAP alone, in preterm neonates with RDS, as assessed by pre-specified outcome measures. In addition, this study will evaluate the device and the ability to administer up to 3 repeat doses.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF from legally authorized representative.
* Gestational age: 26 to 32+6 weeks PMA.
* Successful implementation of non-invasive support or ventilation within 30 minutes after birth.
* Spontaneous breathing.
* Investigator determination of RDS. A chest x-ray should be obtained before treatment to confirm the diagnosis.
* Within the first 6 hours after birth, requires an nCPAP of 5 to 7 cm H2O that is clinically indicated for at least 15 minutes with an FiO2 > 0.25 to ≤ 0.35 to maintain SpO2 of 90% to 95%.

Exclusion Criteria:

* A heart rate that cannot be stabilized above 100 bpm within 5 minutes of birth.
* Recurrent episodes of apnea requiring positive pressure ventilation.
* A 5 minute Apgar score < 5.
* Major congenital malformation(s) or craniofacial abnormalities that preclude the use of nCPAP.
* Clinically significant diseases or conditions other than RDS which could potentially interfere with cardiopulmonary function.
* A known or suspected chromosomal abnormality or syndrome.
* Premature rupture of membranes > 3 weeks.
* Hemodynamic instability requiring vasopressors or steroids for hemodynamic support and/or presumed clinical sepsis.
* A need for intubation and/or invasive mechanical ventilation at any time before enrollment into the study.
* The administration (or plan for administration) of another investigational agent or investigational medical device, any other surfactant agent, or systemic corticosteroids.
* Presence of air leak on the baseline chest radiograph or diagnosed via ultrasound or illumination.

Ages: 30 Minutes to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Guardia, MD, Principal Investigator — Windtree Therapeutics, Inc.
Locations (3):
- Poland (3):
  - Szpital Specjalistyczny nr 2 w Bytomiu Oddzial Noworodkow Blok Va, Bytom
  - Ginekologiczno-Polozniczy Szpital Kliniczny Uniwewersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Samodzielny Publiczny Spcjalistyczny Zaklad Opieki Zdrowotnej "Zdroje", Oddzial Noworodkow, Szczecin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: 18 April 2020 to 19 January 2021 Enrollment occurred in neonatal intensive care units.
Pre-assignment Details: Subjects were screened before enrollment. Screen fail reasons included: unable to maintain required FiO2 (majority of screen fails), no determination of RDS, need for mechanical ventilation, outside of enrollment window
Groups:
- Lucinactant (160 mg/kg) + nCPAP: Lucinactant for inhalation, 160 mg total phospholipids (TPL)/kg Delivered as an aerosol, with up to 3 repeats of 80 mg/kg allowed within 36 hours of birth
  Lucinactant for Inhalation: A drug-device combination product that delivers aerosolized SRT to preterm neonates with RDS who are being supported with nCPAP.
- nCPAP Only: nCPAP Only as sham comparator. Bubble nCPAP is standard of care. Treatment time behind barrier to match active treatment delivery time
  nCPAP Only: Nasal CPAP Alone
Period: Overall Study
Arm/Group | Lucinactant (160 mg/kg) + nCPAP | nCPAP Only
Started | 11 | 1
Completed | 11 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Lucinactant (160 mg/kg) + nCPAP | nCPAP Only | Total
Number analyzed (Participants) | 11 | 1 | 12
Age, Continuous [Median (Full Range); unit: hours] — Subjects are newborns
  hours | 3.25 [1.05 to 4.85] | 1.05 [1.05 to 1.05] | 3.02 [1.05 to 4.85]
Age, Customized [Median (Inter-Quartile Range); unit: weeks] — Gestational Age (GA) in weeks
  weeks
    Gestational Age | 30.3 [28.4 to 32.6] | 31.0 [31 to 31] | 30.4 [29.1 to 31.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 7 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 1 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 1 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Poland | 11 | 1 | 12
Apgar Score at One Minute [Median (Full Range); unit: Scores on a scale] — Apgar score measures appearance, pulse, grimace, activity, and respiration. Scores range from 0 to 10 (0 to 2 for each component with 2 being the best). A score of 7-10 is considered "reassuring." Measured at 1 or 5 minutes after birth for this study.
  Scores on a scale | 7.0 [4 to 9] | 7.0 [7 to 7] | 7.0 [4 to 9]
Apgar Score at Five Minutes [Median (Full Range); unit: Scores on a scale] — Apgar score measures appearance, pulse, grimace, activity, and respiration. Scores range from 0 to 10 (0 to 2 for each component with 2 being the best). A score of 7-10 is considered "reassuring." Measured at 1 or 5 minutes after birth for this study.
  Scores on a scale | 8.0 [7 to 8] | 8.0 [8 to 8] | 8.0 [7 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Failure or Death
Description: Number of participants with respiratory failure due to RDS or death. Respiratory failure due to RDS is defined as intubation for mechanical ventilation and/or surfactant administration
Time Frame: 28 days of life
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Lucinactant (160 mg/kg) + nCPAP | nCPAP Only
Number analyzed (Participants) | 11 | 1
Participants | 6 | 0

2. Secondary Outcome: Number With BPD
Description: Number of participants with bronchopulmonary dysplasia (BPD)
Time Frame: 36 weeks post-menstrual age (PMA)
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Groups:
- Lucinactant (160 mg/kg) + nCPAP: Lucinactant for inhalation, 160 mg total phospholipids (TPL)/kg Delivered as an aerosol once, with up to 3 repeats of 80 mg/kg allowed within 36 hours of birth
  Lucinactant for Inhalation: A drug-device combination product that delivers aerosolized SRT to preterm neonates with RDS who are being supported with nCPAP.
Arm/Group | Lucinactant (160 mg/kg) + nCPAP | nCPAP Only
Number analyzed (Participants) | 11 | 1
Participants | 0 | 0

3. Secondary Outcome: Mortality
Description: All-cause mortality
Time Frame: 36 weeks PMA or 28 days of life (whichever is later)
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Lucinactant (160 mg/kg) + nCPAP | nCPAP Only
Number analyzed (Participants) | 11 | 1
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Common Complications of Prematurity
Description: Number of participants with complications including intraventricular hemorrhage, periventricular leukomalacia, pulmonary hemorrhage, apnea, necrotizing enterocolitis, patent ductus arteriosus, acquired sepsis, and retinopathy of prematurity.
Time Frame: 36 weeks PMA
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Lucinactant (160 mg/kg) + nCPAP | nCPAP Only
Number analyzed (Participants) | 11 | 1
Participants | 9 | 1

ADVERSE EVENTS:
Time Frame: Through 36 weeks PMA or discharge/transfer, an average of 28 days of life.
Arm/Group | Lucinactant (160 mg/kg) + nCPAP | nCPAP Only
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/1
Other Adverse Events (participants affected / at risk) | 11/11 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lucinactant (160 mg/kg) + nCPAP (N=11) | nCPAP Only (N=1)
Duodenal atresia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — Worsening congenital partial duodenal artesia
Pneumonediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lucinactant (160 mg/kg) + nCPAP (N=11) | nCPAP Only (N=1)
Anemia neonatal (Blood and lymphatic system disorders) | 8 (9) | 0 (0)
Coagulation disorder neonatal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Congenital pneumonia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Duodenal atresia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotizing enterocolitis neonatal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 3 (3) | 1 (1)
Infusion site extravasation (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Gastric residual assessment (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 7 (8) | 1 (1)
Feeding intolerance (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Osteopenia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation neonatal (Pregnancy, puerperium and perinatal conditions) | 5 (6) | 1 (1)
Bradycardia neonatal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 7 (8) | 0 (0)
Neonatal respiratory distress syndrome (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemostatsis (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiovascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Haemangioma (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early leading to a very small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The preparation and submittal for publication of a manuscript containing the study results shall be in accordance with a process determined by a mutual written agreement among Windtree and participating institutions. The publication or presentation of any study results shall comply with all applicable privacy laws, including but not limited to HIPAA.

DOCUMENTS (3):
  • Study Protocol (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04264156/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT04264156/SAP_001.pdf
  • Informed Consent Form (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT04264156/ICF_002.pdf